CLINICAL TRIAL: NCT02530983
Title: Mayo Clinic Upper Digestive Disease Survey
Acronym: UDD
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Luis F. Tapias Vargas, Principal Investigator, Mayo Clinic
Other Study IDs: 14-009873
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Neoplasms; Cancer of Esophagus; Cancer of the Esophagus; Esophageal Cancer; Esophagus Cancer; Neoplasm, Esophageal; Esophagectomy; Abnormalities, Digestive System; Digestive System Abnormalities
MeSH Terms: conditions — Esophageal Neoplasms; Digestive System Abnormalities | interventions — Amyloid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Esophagectomy/Esophageal Reconstruction/Treatment: Patients who have undergone esophagectomy, esophageal reconstruction, or treatment
  Interventions: Other: Mayo Clinic Upper Digestive Disease Survey on Paper; Other: Upper Digestive Disease (UDD Monitor) App
- Upper Digestive Disease: Patients who have an upper digestive disease.
  Interventions: Other: Mayo Clinic Upper Digestive Disease Survey on Paper; Other: Upper Digestive Disease (UDD Monitor) App

INTERVENTIONS:
Other: Mayo Clinic Upper Digestive Disease Survey on Paper — Mayo Clinic patients will be asked to complete the Mayo Clinic Upper Digestive Disease Survey at their one month surgical follow up visit and then every three months for 1 year after surgery, then with each surveillance clinic visit or a minimum of once per year for their lifetime. The questionnaire can be completed at their clinic visit, over the telephone, or by mail. The patient's medical record will also be reviewed to gather any other contributing information.
Other: Upper Digestive Disease (UDD Monitor) App — Mayo Clinic and non Mayo Clinic patients can participate by loading the app through the app store. Patient consent will be completed in the app. Patients will be asked to complete questionnaires at their 1.5 month surgical or diagnosis follow up and then every three months for 1 year after their surgery or diagnosis, then with each surveillance clinic visit or a minimum of once per year for their lifetime or as long as they want to participate.
  for iOS: https://apps.apple.com/us/app/upper-digestive-disease/id6448756724 for Android: https://play.google.com/store/apps/details?id=com.mayoclinic.uddmobile&pli=1

SUMMARY:
The Mayo Clinic Conduit Report Card Questionnaires have been created in order to have a consistent evaluation tools for patients undergoing esophageal reconstruction or treatment or patients that are experiencing an upper digestive disease in order to standardize and validate outcome measures. Data will be used to establish the validation of the questionnaires/survey. Data will also lead to the establishment of "normal" or expected scores for patients undergoing each type of esophagectomy procedure and for upper digestive diseases. Data will contribute to creating treatment algorithms for symptom management for upper digestive diseases and for post-operative complications and symptoms as well as contribute to pre-operative education.

DETAILED DESCRIPTION:
The Mayo Clinic Conduit Report Card Questionnaires are a compilation of standard questionnaires and questions that have been created specifically for this study some of which are patient report and others that are administered by the provider or study staff. It includes the Promis Global Health Score, modified Mayo GER Score questions, modified Dysphagia Questionnaire-30 Day questions, and Zubrod Score. It also includes a 10-point scale to grade postoperative pain, milk assessment, Modified Mayo Reflux Score adapted from the Mayo Clinic Reflux Score, Dumping Score adapted from Sigstad's Scoring System, Simple Dysphagia Score adapted from Mellows and Pinkas, Stricture Score adapted from Blackmon, et al., Pyloric Spasm Score, and Conduit Emptying Score abstracted from Vaezi, Baker, Achkar, and Richter. We will also be collecting information on their demographics, operation, nutritional status, laboratory values, testing results and clinical outcomes.

Patients will be asked to complete the Mayo Clinic Upper Digestive Disease Survey at their one month surgical follow up visit and then every three months for 1 year after surgery, then with each surveillance clinic visit or a minimum of once per year for their lifetime for patients who undergo surgery and at one month following diagnosis and then every three months for 1 year after diagnosis, then with each surveillance clinic visit or a minimum of once per year for their lifetime for patients that do not undergo surgery. The questionnaire can be completed at their clinic visit, over the telephone, or by mail using the paper form or may be completed using an electronic application. The electronic version is available for Mayo Clinic and non Mayo Clinic patients through the app store in conjunction Mayo IT.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing or having already undergone an esophagectomy or esophageal reconstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing or having already undergone an esophagectomy or esophageal reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Completion of the Mayo Clinic Upper Digestive Disease Survey by patients at varying time points following surgery | 1 year
  Completed Mayo Clinic Upper Digestive Disease Survey will be analyzed and used to establish validation.

SECONDARY OUTCOMES:
Establishment of "normal" or expected scores from the Mayo Clinic Upper Digestive Disease Survey | 3 years
  Completed Mayo Clinic Upper Digestive Disease Survey will be used in the establishment of "normal" or expected scores for patients undergoing each type of esophagectomy procedure at different time points following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Tapias Vargas, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No